CLINICAL TRIAL: NCT01674088
Title: The Use of a Novel 13C Sucrose Breath Test (13C SBT) to Determine Intestinal Permeability in Irritable Bowel Syndrome (IBS) Patients
Brief Title: Sucrose Breath Test to Determine Intestinal Permeability in IBS
Status: Completed | Type: Observational
Sponsor: Metabolic Solutions Inc. (Industry)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: SBT-01
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; breath testing; carbon-13
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Irritable Bowel Syndrome: Subjects meeting Rome III criteria will be included as the group Irritable Bowel Syndrome
- Healthy Controls: Subjects not meeting Rome III criteria and meeting clinical definitions of general good health will be considered as Healthy Controls

SUMMARY:
Irritable Bowel Syndrome (IBS) is a growing clinical diagnosis affecting 10-20% of the US population. While current diagnostic criteria aids in correctly diagnosing IBS, the cause of the disease still remains unclear. It has been hypothesized that patients with IBS have alterations in the intestinal lining leading to release of toxic substances into the blood, commonly referred to as leaky gut. Current methods used to study leaky gut are both expensive and invasive. The investigators will test a new breath test to measure leaky gut in both IBS patients and subjects without IBS symptoms.

DETAILED DESCRIPTION:
The sucrose breath test involves taking by mouth 20 grams of common sucrose. This amount of sucrose is about 4 packets of sugar that you would use to sweeten a beverage. If subjects meet eligibility criteria, a single breath test will be conducted on all subjects. The breath test involves collecting breath by exhaling through a straw into a special test tube. A breath sample is collected before administration of sucrose. After the baseline breath sample, a sugar solution with the 20 grams of sucrose is administered by mouth. Three additional breath samples are collected at 30, 60 and 90 minutes. After 90 minutes, the protocol is finished. We will be analyzing breath carbon dioxide for different levels of heavy carbon atoms (carbon-13)with an instrument called an isotope ratio mass spectrometer. Our study plan is to compare the amount of carbon-13 in breath between IBS patients and subjects without the condition. Up to 20 subjects per group will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Male or females with clinical diagnosis of Irritable Bowel Syndrome by Rome III criteria (IBS Group) or healthy control.
* Must be 18 years old or greater.
* Women of child-bearing potential must have a negative pregnancy test.

Exclusion Criteria:

* Females who are lactating or pregnant.
* Subjects with allergy to sucrose.
* Subjects with other causes of abdominal pain or altered bowel habits such as IBD, celiac disease, pancreatitis or gastrointestinal bleeding.
* Subjects with a history of diabetes mellitus.
* Subjects with a recent febrile illness (5 days prior to study).
* Subjects that received an investigational drug or device within 30 days prior to study entry.
* Subjects that do not have the mental capacity to understand the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinics of Shands Hospital, Gainesville, FL, residents within Gainesville, FL and students of the University of Florida.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Area under the breath 13CO2 concentration versus time curve (AUC) of sucrose | 90 minutes
  AUC curves will be generated after measurement of breath carbon-13 labeled carbon dioxide over 90 minutes of collection.

CONTACTS AND LOCATIONS:
Overall Officials: David A Wagner, PhD, Principal Investigator — Metabolic Solutions Inc.
Locations (1):
- University of Florida Shands Hospital, Gainesville, Florida, United States